CLINICAL TRIAL: NCT05798949
Title: Chronic Pain Rehabilitation in Patients With Small Fiber Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Catharina G. Faber, Professor, Academisch Ziekenhuis Maastricht
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SFN-rehabilitation
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Sequential replicated randomized single-case experimental-design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure in vivo-therapy (Active Comparator): In the first phase, patients with idiopathic small fiber neuropathy will receive exposure in vivo therapy for at least 4 weeks, 2 sessions/week.
  In the second phase, the therapy will be expanded with either 4 weeks or 6 weeks, 2sessions/week, depending on the outcome of the first session.
  Interventions: Behavioral: Chronic pain rehabilitation: exposure in vivo
- Graded activity-therapy (Active Comparator): In the first phase, patients with idiopathic small fiber neuropathy will receive graded activity-therapy for at least 4 weeks, 2 sessions/week.
  In the second phase, the therapy will be expanded with either 4 weeks or 6 weeks, 2sessions/week, depending on the outcome of the first session.
  Interventions: Behavioral: Chronic pain rehabilitation: graded activity
- Acceptance and commitment therapy (Active Comparator): In the first phase, patients with idiopathic small fiber neuropathy will receive acceptance and commitment therapy for at least 4 weeks, 2 sessions/week.
  In the second phase, the therapy will be expanded with either 4 weeks or 6 weeks, 2sessions/week, depending on the outcome of the first session.
  Interventions: Behavioral: Chronic pain rehabilitation: acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Chronic pain rehabilitation: exposure in vivo — Behavioral, chronic pain rehabilitation therapy
  Other Names: Exposure in vivo
  Arms: Exposure in vivo-therapy
Behavioral: Chronic pain rehabilitation: graded activity — Behavioral, chronic pain rehabilitation therapy
  Other Names: graded activity
  Arms: Graded activity-therapy
Behavioral: Chronic pain rehabilitation: acceptance and commitment therapy — Behavioral, chronic pain rehabilitation therapy
  Other Names: acceptance and commitment therapy
  Arms: Acceptance and commitment therapy

SUMMARY:
Small fiber neuropathy (SFN) is a condition that is dominated by invalidating neuropathic pain. Pharmacological neuropathic pain treatment is often disappointing, since pain reduction is mostly slight and side effects can be debilitating. Although neuropathic pain is caused by a lesion of the somatosensory system, also psychological factors, such as fear and catastrophizing, appear to play a role in the origin and maintenance of disability in chronic pain. Rehabilitation based on pain education and cognitive behavioral treatment including elements of acceptance and commitment therapy, exposure in vivo or graded activity can be performed to influence these factors. To date no specific rehabilitation programs are available for patients diagnosed with SFN.

DETAILED DESCRIPTION:
Small fiber neuropathy (SFN) presents with neuropathic pain and autonomic dysfunction, caused by damage of the myelinated Aδ- and unmyelinated C-fibers. Neuropathic pain in SFN is chronic and severe. In 47% of the SFN cases, an underlying cause can be found. The diagnosis of SFN is established on the clinical signs and symptoms, in combination with reduced intra-epidermal nerve fiber density in the skin biopsy and/or abnormal quantitative sensory testing, with no abnormalities in the nerve conduction test (no large fiber involvement). Without underlying cause or when causative treatment is not sufficient, the treatment is focused on symptomatic neuropathic pain relief. Nevertheless, current pharmacological treatment is not sufficient enough in pain relief. In less than 50% of the pain patients, pain reduction of 30-40% has been observed with the most potent analgesia. Besides the lack of effectiveness of pharmacological medication, side effects and abuse are reported. These insufficient treatment options of SFN enables the necessity to search for other possible treatments.

In the treatment of (chronic) pain disability, a biopsychosocial approach seems to be effective in reducing disability and quality of life (QOL) in SFN. As we know based on earlier studies, chronic (neuropathic) pain, such as SFN, is influenced by several psychological factors, especially in causing and perpetuating pain. First, catastrophizing is one of those disabling psychological factors, which is defined as exaggerated negative mental set brought to bear during actual or anticipated pain experience Catastrophizing is seen as a precursor of pain, rather than consequence. Evidence showed a relation between the severity of chronic neuropathic pain and catastrophizing. Pain catastrophizing has been correlated to pain intensity, independent of physical impairment. In chronic pain, negative and catastrophic thoughts about illness often increase the level of disability. It seems that catastrophizing is one of the factors influencing QOL. Second, fear is another disabling psychological factor. Fear of pain can result in avoidance behavior and reduction of daily activities. Avoidance is the behavior aimed at postponing or preventing an aversive situation from occurring, which are mostly seen as a threat. According to the basic fear avoidance (conditioning) model, chronic pain and disability are induced by behavior. Neutral stimulus receives a negative load. In daily activities, these stimuli will remind patients to the painful experiences and so predicting pain. The intensity of pain combined with psychosocial factors can result in escape and avoidance behavior with eventually an impact for the level of physical activity.

These factors can be treated with cognitive behavioral therapy (CBT), which aims to change the behavior, mindset, or feelings of the patient, helping to experience less distress, enjoying more and being more productive. Varying CBT modalities exists: exposure in vivo, acceptance and commitment therapy (ACT), and graded activity (GA), which will be discussed. All the mentioned modalities will be provided by a treatment team consisting of a psychologist and an occupational therapist, whom both are experienced in the modalities of CBT. For every patient an individualized program will be designed based on the results of a screening. First, a patient will receive education about disabling factors that interfere with functioning in their personal situation. Thereafter, an individual treatment plan containing elements that specifically target disabling factors in the patient's situation will guide further treatment. Additional treatment elements can be based on three cognitive behavioral approaches: exposure in vivo, graded activity and acceptance commitment therapy (ACT). One or more modalities can be combined.

The main (primary) objective is to test the effectiveness of a personally tailored rehabilitation treatment targeting the specific psychological and behavioral factors related to decreasing disability, and improving QOL in SFN. The secondary objective is the personally tailored rehabilitation treatment program will have decrease of pain intensity, mood, and pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

* Aged older than 18 years,
* Skin-biopsy proven idiopathic small fiber neuropathy (SFN),
* Main goal/purpose to achieve with rehabilitation therapy.

Exclusion Criteria:

* Are not able to provide written informed consent,
* Have an underlying condition of SFN (diabetes, SCN (sodium voltage-gated channel alpha) 9A (subunit 9A) /10A (subunit 10A) /11A (subunit 11A) mutation, hypothyroidism, renal failure, vitamin B12 deficiency, monoclonal gammopathy of undetermined significance, alcohol abuses, malignancies, chemotherapeutic drugs),
* Have other neurological disease than SFN that may cause pain in the feet and/or damage to the somatosensory nervous system, are excluded,
* Have received any form of cognitive behavioral therapy within the last 6 months will be excluded from this study,
* Have insufficient comprehension of the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Disability measured with small fiber neuropathy rash built overall disability scale (SFN-RODS) | Through study completion, an average of 1 year
  This is a questionnaire consisting of 12 questions, in which a higher score is indicating more disability. There is no cut-off point. The minimum score is 0. The maximum score is 100.
Health related quality of life measured with short form 12 questionnaire (SF-12) | Through study completion, an average of 1 year
  This is a questionnaire consisting of 8 items measuring the quality of life, in which a lower score is indicating a lower quality of life compared to healthy individuals. The minimum score is 0, and the maximum score is 100.

SECONDARY OUTCOMES:
Pain intensity measured with numeric rating scale (NRS) | Through study completion, an average of 1 year
  This is a measurement about the pain intensity. On a scale of 0-10 (Likert 11), a higher score is indicating more pain, in which 0 is indicating no pain at all (minimum score), and 10 is indicating the worst pain ever. (maximum score).
Mood measured with hospital anxiety and depression scale (HADS) | Through study completion, an average of 1 year
  HADS is a questionnaire measuring symptoms of anxiety and depression with 14 questions, consisting of 2 subscales (with each 7 items): a score between 0-7 is seen as normal, between 8-10 is seen as borderline, and a score higher than 11 indicates an underlying anxiety or depressive disorder. The minimum score is 0, and the maximum score is 21.
Pain catastrophizing measured with pain catastrophizing scale (PCS) | Through study completion, an average of 1 year
  PCS is a questionnaire consisting of 13 questions, a higher score is indicating the presence of more catastrophic thoughts, there is no cut-off point. The minimum score is 0, and the maximum score is 52.

CONTACTS AND LOCATIONS:
Overall Officials: J. AC Verbunt, MD, PhD, Principal Investigator — Adelante Zorggroep; J. GJ Hoeijmakers, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Adelante Zorggroep, Maastricht, Limburg
  - Maastricht University Medical Center, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damci A, den Hollander M, Hoeijmakers JGJ, Faber CG, Goossens MEJB, Verbunt JAMCF. Biopsychosocial rehabilitation therapy in small fiber neuropathy: research protocol to study the effect of rehabilitation treatment. Front Neurol. 2024 Nov 13;15:1493326. doi: 10.3389/fneur.2024.1493326. eCollection 2024. PMID 39606707